CLINICAL TRIAL: NCT04769609
Title: Reconstructive Surgical Therapy of Peri-implantitis: 3-year Results of a Randomized Clinical Trial
Brief Title: Reconstructive Surgical Therapy of Peri-implantitis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Assoc. Professor, Gazi University
Other Study IDs: GUDHKAEK.2021.01/4
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; biomaterials; surgical treatment
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concentrated growth factor (CGF) group: Reconstructive surgical therapy of peri-implantitis using a bone substitute combined with CGF
  Interventions: Device: bioresorbable membrane
- Collagen membrane (CM) group: Reconstructive surgical therapy of peri-implantitis using a bone substitute combined with CM
  Interventions: Device: bioresorbable membrane

INTERVENTIONS:
Device: bioresorbable membrane — reconstructive surgical treatment of peri-implant bone defects

SUMMARY:
Various treatment protocols of peri-implantitis involving surgical therapies with open flap debridement procedures, resective or reconstructive modalities have been documented to achieve variable success. Surgical non-reconstructive approaches have been suggested to have limited effectiveness in terms of the resolution of inflammation in the long term. Therefore, much more interest has been intensified regarding the efficacy of biomaterials used in reconstructive approaches. The aim of this study was to investigate the 3-year clinical/radiographic outcomes of reconstructive surgical therapy of peri-implantitis using a bone substitute combined with two different bioresorbable barrier membranes, either collagen membrane (CM) or concentrated growth factor (CGF). A total of 52 patients who had at least one implant diagnosed with peri-implantitis and needed to be scheduled for reconstructive therapy of a peri-implant infrabony defect were included. Peri-implantitis case was defined as increased probing depth (PD) compared to previous examinations with bleeding on probing (BOP) and/or suppuration and radiographic evidence of peri-implant bone loss beyond crestal bone level changes resulting from initial bone remodeling. The patients were randomly assigned to receive a bone substitute filling in combination with either CM or CGF. Intrabony components were filled with a bone substitute (BioOss spongiosa granules; Geistlich, Wolhusen, Switzerland) and covered with a CM (Bio-Guide, Geistlich Biomaterials) or CGF membrane. The plaque index (PI), gingival index (GI), BOP, PD, clinical attachment level (CAL), mucosal recession (MR) and radiographic vertical defect depth (VDD) values were evaluated at 1 and 3 years postoperatively.

DETAILED DESCRIPTION:
Peri-implantitis is a plaque-associated pathological disease affecting the soft and/or hard tissues surrounding a dental implant and clinically characterized by bleeding on probing (BOP) and/or suppuration (Supp), increased probing depths (PDs) and/or mucosal marginal recessions (MRs) in addition to radiographic marginal bone loss (MBL) compared to previous examinations. Considering the increasing numbers of patients undergoing restorative treatment through dental implants and the corresponding increase in the prevalence of peri-implantitis, it is imperative to perform effective treatment methods for the management of these conditions. On the basis of evidence, the most reliable and predictable treatment of peri-implantitis has not yet been described, moreover, if the disease is left untreated, it progresses in a non-linear accelerating manner. Hence, peri-implantitis has been considered to be a major, unpredictable and growing problem for clinicians.

Various treatment protocols of this challenging problem involving non-surgical approaches and surgical therapies with open flap debridement procedures, resective surgeries, or reconstructive modalities, which include the use of bone substitutes with or without a membrane, decontamination methods of implant surfaces, antimicrobial prescriptions whether to use submerged or non-submerged techniques, have been proposed. Although non-surgical interventions have been reported to be effective in reducing BOP and PDs in peri-implantitis sites, these therapies have appeared to be unpredictable for the management of peri-implantitis, especially in most severe cases. As another treatment option, surgical non-reconstructive approaches, i.e. open flap debridement and surface decontamination alone, have been suggested to have limited effectiveness in terms of the resolution of inflammation for the long-term outcomes. Therefore, much more interest has been intensified regarding the efficacy of biomaterials used in reconstructive approaches. Several surgical augmentative therapy studies, including the use of bone substitutes with or without barrier membranes have demonstrated significant clinical and radiographic improvements for at least 3 years, especially in well-contained (three- or four-wall) intrabony defects. A systematic review evaluating long-term outcomes of reconstructive therapy for the management of peri-implantitis showed a mean PD reduction of 3 mm and a radiographic gain of 2.4 mm in bone level. However, as indicated by the last EFP Workshop, no evidence to support the superiority of a specific material, product or membrane in terms of long-term clinical outcomes of a reconstructive approach has been found. It has been strictly recommended that identification of peri-implantitis therapy success and disease resolution in the long-term management are required to allow adequate assessment of stable treatment outcomes.

Because of many studies indicating that growth factors have provided to transiently stimulate cells locally, accelerate angiogenesis, promote proliferation, differentiation, and regeneration, the additional use of them in the management of peri-implantitis has been proposed to improve the clinical outcomes and enhance soft and hard tissue regeneration. A recent systematic review and meta-analysis has been suggested that growth factors might be associated with better outcomes with regard to PD and BOP, whereas, they did not reveal statistically significant evidence for yielding additional benefits in the treatment of peri-implantitis. A randomized clinical trial (RCT) on the reconstructive surgical treatment of peri-implantitis evaluating concentrated growth factor (CGF) used as a bioresorbable barrier membrane in combination with a bone substitute, was performed recently by our study group and demonstrated significant improvements in both clinical and radiographic assessments at 1-year follow-up. Nevertheless, there is scarce information in the literature regarding the predictability and long-term stability of autologous growth factors in peri-implantitis management.

It is, therefore, the aim of this study to investigate the 3-year clinical/radiographic outcomes of reconstructive surgical therapy of peri-implantitis using a bone substitute combined with two different bioresorbable barrier membranes, either collagen membrane (CM) or CGF, and moreover, to identify prognostic indicators influencing the long-term reconstructive surgical treatment outcome using a multilevel statistical model.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* having at least one implant demonstrating two- or three-wall infrabony defect ≥3 mm, which presented a probing depth of ≥5 mm with BOP and/or suppuration,
* no implant mobility and no evidence of occlusal overload.

Exclusion Criteria:

* serious systemic diseases, medications or conditions that would contraindicate for periodontal surgery and compromise wound healing,
* a history of taking systemic antibiotic during the past 3 months, and
* placement, and prosthetic loading of implants within the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Presence of bleeding on probing (BOP) and/or suppuration (SUP) on gentle probing, and a radiographic marginal bone loss (MBL) ≥ 2 mm based on baseline radiographs taken at the time of prosthesis delivery with increased probing depth (PD) compared to previous examinations.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
mean vertical radiographic defect depth (VDD) | Postoperative 3 years
  Radiographic vertical defect depth (VDD) was measured between the first bone-to-implant contact and the reference point at the coronal part of the implant body at both mesial and distal aspects of the implants.

SECONDARY OUTCOMES:
Plaque index | Baseline, postoperative 1 and 3 years
  Silness & Löe plaque index (PI) marked with a score from 0 to 3 (0: absence of microbial plaque; 1: thin film of microbial plaque; 2: moderate accumulation with plaque in the sulcus; 3: large amount of plaque in sulcus or pocket along the free gingival margin)
Gingival index | Baseline, postoperative 1 and 3 years
  Löe & Silness index (GI) marked with a score from 0 to 3. (0: normal gingiva; 1: mild inflammation, 2: moderate inflammation, 3: severe inflammation)
Bleeding on probing (percent [%]) (BOP) | Baseline, postoperative 1 and 3 years
  BOP was assessed according to presence or absence of bleeding 30 s after gentle probing
Probing depth (mm) (PD) | Baseline, postoperative 1 and 3 years
  PD was measured as the distance from the mucosal margin to the bottom of the probeable pocket
Clinical attachment level (mm) (CAL) | Baseline, postoperative 1 and 3 years
  Clinical attachment level (CAL) defined as PD+ mucosal recession.
Mucosal recession (mm) (MR) | Baseline, postoperative 1 and 3 years
  Mucosal recession (MR) was measured as the distance from the mucosal margin and the implant abutment interface

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Result] Mercado F, Hamlet S, Ivanovski S. Regenerative surgical therapy for peri-implantitis using deproteinized bovine bone mineral with 10% collagen, enamel matrix derivative and Doxycycline-A prospective 3-year cohort study. Clin Oral Implants Res. 2018 Jun;29(6):583-591. doi: 10.1111/clr.13256. Epub 2018 May 16. PMID 29767434
- [Result] La Monaca G, Pranno N, Annibali S, Cristalli MP, Polimeni A. Clinical and radiographic outcomes of a surgical reconstructive approach in the treatment of peri-implantitis lesions: A 5-year prospective case series. Clin Oral Implants Res. 2018 Oct;29(10):1025-1037. doi: 10.1111/clr.13369. Epub 2018 Sep 28. PMID 30267445
- [Result] Tomasi C, Regidor E, Ortiz-Vigon A, Derks J. Efficacy of reconstructive surgical therapy at peri-implantitis-related bone defects. A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:340-356. doi: 10.1111/jcpe.13070. PMID 30667523
- [Result] Polymeri A, Anssari-Moin D, van der Horst J, Wismeijer D, Laine ML, Loos BG. Surgical treatment of peri-implantitis defects with two different xenograft granules: A randomized clinical pilot study. Clin Oral Implants Res. 2020 Nov;31(11):1047-1060. doi: 10.1111/clr.13651. Epub 2020 Sep 9. PMID 32803798
- [Result] Renvert S, Roos-Jansaker AM, Persson GR. Surgical treatment of peri-implantitis lesions with or without the use of a bone substitute-a randomized clinical trial. J Clin Periodontol. 2018 Oct;45(10):1266-1274. doi: 10.1111/jcpe.12986. Epub 2018 Aug 21. PMID 30003583
- [Result] Roccuzzo M, Layton DM, Roccuzzo A, Heitz-Mayfield LJ. Clinical outcomes of peri-implantitis treatment and supportive care: A systematic review. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:331-350. doi: 10.1111/clr.13287. PMID 30328195
- [Result] Isehed C, Svenson B, Lundberg P, Holmlund A. Surgical treatment of peri-implantitis using enamel matrix derivative, an RCT: 3- and 5-year follow-up. J Clin Periodontol. 2018 Jun;45(6):744-753. doi: 10.1111/jcpe.12894. Epub 2018 Apr 26. PMID 29574866
- [Result] Khoury F, Keeve PL, Ramanauskaite A, Schwarz F, Koo KT, Sculean A, Romanos G. Surgical treatment of peri-implantitis - Consensus report of working group 4. Int Dent J. 2019 Sep;69 Suppl 2(Suppl 2):18-22. doi: 10.1111/idj.12505. PMID 31478576
- [Result] Roccuzzo M, Fierravanti L, Pittoni D, Dalmasso P, Roccuzzo A. Implant survival after surgical treatment of peri-implantitis lesions by means of deproteinized bovine bone mineral with 10% collagen: 10-year results from a prospective study. Clin Oral Implants Res. 2020 Aug;31(8):768-776. doi: 10.1111/clr.13628. Epub 2020 Jul 24. PMID 32559322
- [Result] Monje A, Pons R, Roccuzzo A, Salvi GE, Nart J. Reconstructive therapy for the management of peri-implantitis via submerged guided bone regeneration: A prospective case series. Clin Implant Dent Relat Res. 2020 Jun;22(3):342-350. doi: 10.1111/cid.12913. Epub 2020 May 14. PMID 32410379
- [Result] Aghazadeh A, Persson RG, Renvert S. Impact of bone defect morphology on the outcome of reconstructive treatment of peri-implantitis. Int J Implant Dent. 2020 Jun 17;6(1):33. doi: 10.1186/s40729-020-00219-5. PMID 32548733
- [Result] Carcuac O, Derks J, Abrahamsson I, Wennstrom JL, Petzold M, Berglundh T. Surgical treatment of peri-implantitis: 3-year results from a randomized controlled clinical trial. J Clin Periodontol. 2017 Dec;44(12):1294-1303. doi: 10.1111/jcpe.12813. Epub 2017 Nov 10. PMID 28902426
- [Result] Khouly I, Pardinas-Lopez S, Ruff RR, Strauss FJ. Efficacy of growth factors for the treatment of peri-implant diseases: a systematic review and meta-analysis. Clin Oral Investig. 2020 Jul;24(7):2141-2161. doi: 10.1007/s00784-020-03240-5. Epub 2020 May 16. PMID 32418012
- [Derived] Isler SC, Soysal F, Ceyhanli T, Bakirarar B, Unsal B. Efficacy of concentrated growth factor versus collagen membrane in reconstructive surgical therapy of peri-implantitis: 3-year results of a randomized clinical trial. Clin Oral Investig. 2022 Aug;26(8):5247-5260. doi: 10.1007/s00784-022-04493-y. Epub 2022 May 26. PMID 35618961